CLINICAL TRIAL: NCT00608959
Title: A Single- Center, Open-Label, Study of the Persistence of Antimicrobial Activity of Omiganan 1% Gel vs. Chlorhexidine 2% for Topical Skin Antisepsis in Healthy Adult Subjects
Brief Title: Study of Antimicrobial Activity of Omiganan 1% Gel vs. Chlorhexidine 2% for Topical Skin Antisepsis in Healthy Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cadence Pharmaceuticals (Industry)
Responsible Party: Catherine Hardalo, MD. Vice President, Anti Infectives Clinical Development, Cadence Pharmaceuticals,Inc.
Organization: Cadence (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPI-226-301
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2010-01-25 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Infection
Keywords: Skin colonization; Catheter colonization; Catheter site infection
MeSH Terms: conditions — Infections | interventions — Omiganan; Gels; Chlorhexidine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- omiganan 1% gel (Experimental): Omiganan has a rapid bactericidal and fungicidal effect which is under development for the prevention of infections arising from short-term central venous catheters, as well as for the prevention of surgical wound infections in contaminated wounds.
  Interventions: Drug: omiganan 1% gel
- chlorhexidine 2% (Active Comparator)
  Interventions: Drug: chlorhexidine 2% solution

INTERVENTIONS:
Drug: omiganan 1% gel — Omiganan 1% gel will be applied to 6 sites on the chest and/or abdomen.Swab cultures will be obtained at specified timepoints over a period of 3 days (Part1) or 7 days (Part 2).
  In addition, subjects in Part 2 will have omiganan 1% gel applied to one intravenous (IV) catheter site.
  Arms: omiganan 1% gel
Drug: chlorhexidine 2% solution — Part 1- chlorhexidine 2% solution will be applied to 6 sites on the chest and/or abdomen. All application sites will be covered with semi-transparent dressings.Swab cultures will be obtained at specific timepoints over a period of 3 days.
  Part 2: Subjects in Part 2 will have chlorhexidine 2% solution applied to one intravenous (IV) catheter site only.
  Arms: chlorhexidine 2%

SUMMARY:
The purpose of this research study is to determine if omiganan 1% gel (the investigational medication in this research study) is effective and safe when compared to chlorhexidine 2% (an FDA approved medication) for killing bacteria (germs) that live on the surface of the skin. Both of the study medications are applied topically (on the surface of the skin).

DETAILED DESCRIPTION:
The study is comprised of 2 parts with approximately 20 subjects participating in each part.

Subjects eligible for Part 1 will have omiganan 1 % gel applied to 6 sites across the chest and/or abdomen and chlorhexidine 2% solution will be applied to 6 matching sites on the contralateral side.

Subjects eligible for Part 2 will each have omiganan 1% gel applied to 6 sites across the upper chest or abdomen.In addition,subjects in Part 2 will have 2 peripheral catheters inserted, one in each arm.One catheter insertion site will be treated with omiganan 1% gel (following treatment with isopropyl alcohol) and the other site will be treated with chlorhexidine 2%/isopropyl alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects18-70 years of age
* No evidence of dermatosis, dermatitis, inflammation, scarring, or acute injuries to the drug application sites on the chest or abdomen
* Subjects must have screening samples from the skin on the right and left side of the chest or abdomen containing at least 2.5 log10 colony forming units per square centimeter (CFU/cm2 )organisms (from the average of 2 samples obtained during screening)
* Willing to provide written informed consent.

Exclusion Criteria:

* Allergies or sensitivities to alcohol, adhesive tape, bandages, latex, chlorhexidine gluconate, or any of the ingredients of omiganan 1% gel
* Prior treatment with any systemic antibiotic, or any other product known to affect the normal microbial flora of the skin within 7 days of the screening examination
* Requirement for topical antibiotic use on or within 10 cm of any study test site
* Subjects who have been treated with any investigational drug (other than omiganan) within the previous 30 days, or who are participating in an investigational drug study at any time during the course of this study
* Subjects who have been previously treated with omiganan and experienced a possibly related adverse event during the study Note: a wash out period of one week is required prior to participation in Part 2 of the study
* A medical condition that the Investigator believes may interfere with the safety of the subject or the intent and conduct of the study Note: this includes conditions such as: severe eczema, psoriasis and/or dermal infections, old scars, insulin dependent diabetes mellitus, severe immunocompromising conditions, HIV infection, or use of medications that would interfere with assessment of study endpoints
* A current or recent history of illicit drug or alcohol abuse
* Subjects not willing or able to fulfill protocol requirements
* Pregnancy. Women of childbearing potential who have a positive or equivocal result on a urine and/or blood pregnancy test before study enrollment will not be included

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Hardalo, MD, Study Director — Cadence Pharmaceuticals
Locations (1):
- BioSciences Lab, Bozeman, Montana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single center in the US, from 12 May 2008 - 03 June 2008. Subjects who participated in Part 1 were allowed to participate in Part 2 after a one week washout period.Subjects were not required to participate in both Parts 1 and 2 of the study.
Pre-assignment Details: Subjects required screening skin samples ( from an average of 2 samples) containing at least 2.5log10 colony forming units per cm2 (CFU/cm2)
Groups:
- Omiganan 1% Gel and Chlorhexidine: In Part 1 each subject had omiganan 1% gel applied to 6 sites located across the chest and/or abdomen and chlorhexidine applied to 6 matching sites on the contralateral side.Swab cultures were taken at specified timepoints over 72 hours.
  In Part 2 each subject had omiganan 1% gel applied to 6 sites across the chest and/or abdomen.Swab cultures were taken at specified timepoints over 7 days.In addition subjects in Part 2 had 2 intravenous (IV) catheters inserted, with one catheter insertion site treated with isopropyl alcohol (prior to insertion) and omiganan 1% gel was applied. Catheter tip samples were taken at pre-specified timepoints over the 7 day period.
Period: Part 1
Arm/Group | Omiganan 1% Gel and Chlorhexidine
Started | 25 (25 subjects each participated in Parts 1 and 2 .A total of 20 subjects participated in both parts.)
Completed | 24
Not Completed | 1
Not completed — Did not meet eligibility criteria | 1
Period: Part 2
Arm/Group | Omiganan 1% Gel and Chlorhexidine
Started | 25 (20 Part 1 subjects also participated in Part 2.Five more subjects were enrolled for a total of 25.)
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Omiganan 1% Gel (Part 2): 25 subjects were treated with omiganan 1% gel at skin and intravenous (IV) sites in Part 2.
- Chlorhexidine 2% (CHG) / Omiganan 1% Gel(Part 1): 25 subjects were treated with chlorhexidine 2% and omiganan 1% in Part 1.
- Total: Total of all reporting groups
Arm/Group | Omiganan 1% Gel (Part 2) | Chlorhexidine 2% (CHG) / Omiganan 1% Gel(Part 1) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 24 | 24 | 48.0
  >=65 years | 1 | 1 | 2.0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.6 (15.13) | 36.6 (15.13) | 38.6 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25.0
  Male | 13 | 12 | 25.0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50.0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Skin Bacterial Counts From Baseline to 72 Hours
Description: Change in the mean number of skin bacterial counts (CFU/cm2) which was calculated by subtracting log10 CFU/cm2 at 72 hours (single sample per subject per timepoint) from the log10 CFU/cm2 at 0 hours (baseline) in Part 2.Baseline was calculated by 'pooling' samples from 6 sites adjacent to each timepoint.
Time Frame: Prior to first application (0 hours) to 72 hours post application
Population: ITT set consists of all subjects who received at least one study treatment and had data available at 72 hours.
Measure: Mean (Standard Deviation); unit: log 10 CFU/cm sq
Groups:
- Omiganan 1% Gel (Part 2): Omiganan 1% gel was applied to 6 sites across the chest and/or abdomen. Swab cultures were obtained at specified timepoints over a period of 3 days.
- Chlorhexidine 2%(Part 1): Chlorhexidine 2% solution was applied to 6 sites on the chest and/or abdomen. Swab cultures were obtained at specific timepoints over 3 days.
Arm/Group | Omiganan 1% Gel (Part 2) | Chlorhexidine 2%(Part 1)
Number analyzed (Participants) | 25 | 24
log 10 CFU/cm sq | -1.91 (1.563) | -1.87 (1.656)
Statistical Analysis 1: Comparison: Omiganan 1% Gel (Part 2); Based on a two-sided test at the 5% level of significance, and assuming a SD of 1.3, a sample size of 20 subjects would provide 90% power to detect a mean change of 0.942. No information was available concerning the within-subject variability between the arms; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.91, 95% CI [-2.55 to -1.26], Standard Deviation 1.563
Statistical Analysis 2: Comparison: Chlorhexidine 2%(Part 1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Median Difference (Final Values) = -1.87, 95% CI [-2.57 to -1.17], Standard Deviation 1.656

2. Primary Outcome: Change in Mean Number of Skin Bacterial Counts From Baseline to 7 Days
Description: Change in the mean number of skin bacterial counts (log 10 CFU/cm2)which was calculated by subtracting log10 CFU/cm2 at 7 days (one sample per site per subject per timepoint) from log10CFU/cm2 at 0 hours in Part 2.Baseline was calculated by 'pooling' samples from 6 sites adjacent to each timepoint.
Time Frame: Prior to first application (0 hours) to 7 days post application.
Population: In Part 2 of the study 25 subjects had only omiganan applied to sites across the upper chest or abdomen.Swab cultures were obtained over a period of 7 days at protocol-specified times
Measure: Mean (Standard Deviation); unit: log 10 CFU/sq. cm
Groups:
- Omiganan 1% Gel (Part 2): Omiganan 1% gel was applied to 6 sites across the chest and/or abdomen. Swab cultures were obtained at specified timepoints over a period of 7 days.
Arm/Group | Omiganan 1% Gel (Part 2)
Number analyzed (Participants) | 25
log 10 CFU/sq. cm | -1.44 (1.511)

3. Primary Outcome: Number of Subjects With Significantly Colonized Catheters, Defined as > or = to 15 Colony Forming Units- CFUs)
Description: Roll plate cultures (quantitative) measured CFU on catheter tips after removal up to 7 days after insertion.
Time Frame: Each sampling point and the rate of catheter colonization for each treatment 72 hours to 7 days.
Population: intravenous (IV) catheters were removed for culture from 5 subjects at 72 hours, 10 subjects at 5 days, and 10 subjects at 7 days.
Measure: Number; unit: participants
Groups:
- Omiganan 1% Gel (Part 2): Subjects in Part 2 had 2 intravenous (IV) catheters inserted, with one catheter insertion site treated with isopropyl alcohol (prior to insertion) and omiganan 1% gel was applied. Catheter tip samples were taken at pre-specified timepoints over the 7 day period.
- Chlorhexidine 2%/ Isopropyl Alcohol: Subjects in Part 2 had 2 intravenous (IV) catheters inserted, with one catheter insertion site treated with chlorhexidine/isopropyl alcohol prior to catheter insertion.Catheter tip samples were taken at pre-specified timepoints over the 7 day period.
Arm/Group | Omiganan 1% Gel (Part 2) | Chlorhexidine 2%/ Isopropyl Alcohol
Number analyzed (Participants) | 25 | 24
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Part 1:Baseline (prior to study medication),6 hrs, 24 hrs, 48 hrs, 72 hours after the application of study medication. Part 2: Baseline, 6 hrs, 24 hrs, 48 hrs, 72 hours, 5 days, 7 days after the application of study medication.
Groups:
- Omiganan 1% Gel (Part 1): In Part 1 each subject had omiganan 1% gel applied to 6 sites located across the chest and/or abdomen.
- Chlorhexidine: In Part 1 each subject had chlorhexidine 2% applied to 6 sites located across the chest and/or abdomen. In Part 2 subjects had chlorhexidine 2%/isopropyl alcohol applied to one intravenous (IV) catheter site.
- Omiganan 1% (Part 2): In Part 2 each subject had omiganan 1% gel applied to 6 sites across the chest and/or abdomen.Omiganan 1% gel was applied to one intravenous (IV) catheter site.
Arm/Group | Omiganan 1% Gel (Part 1) | Chlorhexidine | Omiganan 1% (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 7/25 | 8/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Omiganan 1% Gel (Part 1) (N=25) | Chlorhexidine (N=25) | Omiganan 1% (Part 2) (N=25)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Catheter Site Pain (General disorders) | 0/0 (0) | 7 (7) | 7 (7) — IV catheters were inserted in subjects participating in Part 2 only. Part 1 subjects did not have IV catheters.

LIMITATIONS AND CAVEATS:
FDA reviewer noted that there were multiple endpoints that required multiplicity adjustments to control for the overall type I error rate.Based on feedback the 72 hour endpoint was selected for Part 2 as the primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less